CLINICAL TRIAL: NCT01339676
Title: Colecalciferol as an Add-on Treatment to Subcutaneously Administered Interferon-beta-1b for Treatment of MS
Brief Title: Colecalciferol as an Add-on Treatment to Interferon-beta-1b for Treatment of Multiple Sclerosis (MS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Turku (Other)
Responsible Party: Merja Soilu-Hanninen, MD, PhD, docent, neurologist, University of Turku, Department of Neurology, Turku, Finland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-001958-99; EudraCT 2007-001958-99
Record Dates: First submitted 2011-04-19; First posted 2011-04-21 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-04

CONDITIONS: Multiple Sclerosis
Keywords: Vitamin D; Multiple Sclerosis; MRI; Randomised Trial; Finland
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Once weekly treatment with peroral colecalciferol capsules (Dekristol®, Swiss-Caps, Switzerland) containing 20 mg of colecalciferol corresponding to 20000 IU or 0.5 mg of vitamin D
  Interventions: Drug: Colecalciferol
- 2 (Placebo Comparator): Identically appearing once weekly peroral capsules
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: Colecalciferol — Once weekly treatment with peroral colecalciferol capsules (Dekristol®, Swiss-Caps, Switzerland) containing 20 mg of colecalciferol corresponding to 20000 IU or 0.5 mg of vitamin D
  Other Names: Vitamin D
  Arms: 1
Drug: Placebo capsules — Identically appearing once weekly peroral placebo capsules
  Arms: 2

SUMMARY:
This is a multi-centre, double blind, randomised, placebo controlled, parallel group, phase 4 pilot study investigating colecalciferol (vitamin D3) as an add-on treatment to subcutaneously administered interferon-beta-1b in relapsing-remitting multiple sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 55 years
* remitting-relapsing multiple sclerosis according to McDonald criteria who fulfill the reimbursement criteria for interferon-beta and have used interferon-beta-1b for at least one month
* EDSS (expanded disability statsu scale) ≤ 5
* no neutralising antibodies to INFB as measured by indirect MxA test
* prepared and considered to follow the protocol
* using appropriate contraceptive methods (women of childbearing potential)
* has given informed consent

Exclusion Criteria:

* serum calcium >2.6 mmol/L
* serum 25(OH)D2 (kalsidiol) > 85 nmol/L
* presence of primary hyperparathyroidism (serum intact PTH, parathyroid hormone)>65 ng/L)
* pregnancy or unwillingness to use contraception
* alcohol or drug abuse
* use of glucocorticoid treatment other than intravenous methylprednisolone for treatment of relapses
* current use of other immunomodulatory therapy than interferon-beta-1b
* known allergy to cholecalciferol or arachis oil (peanuts)
* therapy with digitalis, calcitonin or active vitamin D3 analogues during the previous 12 months or multivitamins containing vitamin D during previous two weeks preceding study entry
* any condition predisposing to hypercalcaemia (such as any type of cancer)
* sarcoidosis
* nephrolithiasis or renal insufficiency, serum creatinine above 1.5 times the normal upper reference limit
* significant hypertension (Blood Pressure <180/110 mmHg)
* hyperthyroidism, or hypothyroidism in the year before the study began
* a history of nephrolithiasis during the previous five years
* cardiac insufficiency or significant cardiac dysrhythmia
* unstable or advanced ischaemic heart disease
* has suffered a major depression

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2008-03; Primary Completion 2011-05 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Measure: the proportion of patients with P-PTH< 20 ng/l and S-OH(D)2 > 85 nmol/l at 6 and 12 months | one year

SECONDARY OUTCOMES:
Number of Gadolinium-enhancing lesions on T1 and /or new enlarging lesions on Measure: T2/PD based on MRI done 12 months following randomisation compared with the MRI done at the time of randomisation | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Soilu-Hanninen M, Aivo J, Lindstrom BM, Elovaara I, Sumelahti ML, Farkkila M, Tienari P, Atula S, Sarasoja T, Herrala L, Keskinarkaus I, Kruger J, Kallio T, Rocca MA, Filippi M. A randomised, double blind, placebo controlled trial with vitamin D3 as an add on treatment to interferon beta-1b in patients with multiple sclerosis. J Neurol Neurosurg Psychiatry. 2012 May;83(5):565-71. doi: 10.1136/jnnp-2011-301876. Epub 2012 Feb 22. PMID 22362918